CLINICAL TRIAL: NCT03675646
Title: Comparison of Spinal Morphine With Systemic Analgesia After Urologic Surgery
Brief Title: Spinal Morphine for Postoperative Analgesia in Urology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jiri Malek, Assoc. Prof., M.D., Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: malekj3
Record Dates: First submitted 2018-08-23; First posted 2018-09-18 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Pain, Postoperative
Keywords: morphine spinal; prostatectomy; nephrectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Intervention Model Description: Patient elicited for open prostatectomy or open nephrectomy were given intrathecal morphine in normal saline before induction to general anaesthesia (GA) or GA only. After surgery, time to the first opioid request, total opioid consumption during first 24 hours and 48 hours after surgery and opioid side effects were noticed.
Who Masked: Outcomes Assessor
Masking Description: Only ICU personnel was blinded to the method used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine group M (Experimental): Experimental group M were administered preservative-free morphine 250 mcg in 2.5 ml NS intrathecal using 25 G needle in L1/2 - L5/S1 interspaces.
  Interventions: Drug: Morphine
- Control group C (No Intervention): No intervention

INTERVENTIONS:
Drug: Morphine — Intrathecal injection of 250 mcg preservative-free morphine before surgery
  Other Names: No other names
  Arms: Morphine group M

SUMMARY:
The study was performed in urology patients elicited for open prostatectomy or open nephrectomy. Comparison of analgesic effect between group (M) with spinal morphine before general anaesthesia and group without this intervention was measured.

DETAILED DESCRIPTION:
Patients elicited for open prostatectomy or open nephrectomy were randomly divided in 2 groups. Group M were administered preservative-free morphine 250 mcg in 2.5 ml NS intrathecal using 25 G needle in L1/2 - L5/S1 interspaces. Control group (C) were given no intervention. Placebo intrathecal injection in C was not used because of ethical reason. Standard general anaesthesia was used in both groups. After surgery all patients were transferred to urology ICU and were given standard analgesic regimen according to level of pain measured by numeric rating scale (NRS) 0 - 10: NRS > 3 metamizol 1 g IV every 6 h., max. 4 g/24 h., NRS > 3 paracetamol 1g IV every 6 h., max. 4 g/24 h., NRS > 3 lasting 30 min. after administration of previous ones diclofenac 75 mg IM á 12 h., max. 150 mg/24 h., NRS > 4 morphine 10 mg SC á 6 h. Personnel of ICU was blinded to the analgesic method used.

Noticed parameters: pain intensity (NRS), time to NRS ≥ 4, time to the first morphine request, side effects (respiratory rate <8, SpO2<90 %, nausea, vomiting, naloxone administration for SpO2<88 %, itching).

Standard statistical analysis was used, p value < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria

* elicited open prostatectomy or open nephrectomy

Exclusion Criteria

* drug or alcohol dependence
* psychiatric drug use
* ASA classification IV or V
* general contraindication to neuroaxial injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-03-05 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | 48 hours
  Time to the first morphine request during the first two days of ICU stay after surgery (in hours) and total morphine consumption during the first two days of ICU stay (in mg)

SECONDARY OUTCOMES:
Morphine side effects | 48 hours
  respiratory rate <8, SpO2<90 %, nausea, vomiting, naloxone administration for SpO2<88 %, itching

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Malek, M.D., Principal Investigator — 3rd Medical Faculty, Charles University
Locations (1):
- University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No